CLINICAL TRIAL: NCT00773461
Title: A Randomized, Double Blind Study of Safety and Reduction in Signs and Symptoms During Treatment With Tocilizumab Versus Placebo, in Combination With DMARD Therapy, in Patients With Active Rheumatoid Arthritis and Inadequate Response to Current DMARD Therapy
Brief Title: A Study of Tocilizumab in Combination With DMARD Therapy in Patients With Active Rheumatoid Arthritis.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ML21753
Record Dates: First submitted 2008-10-15; First posted 2008-10-16 (Estimated); Results first posted 2016-07-21 (Estimated); Last update posted 2017-08-01 (Actual); Status verified 2017-06

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — tocilizumab

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: tocilizumab [RoActemra/Actemra]
- 2 (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: tocilizumab [RoActemra/Actemra] — 8mg/kg iv every 4 weeks for 24 weeks
  Arms: 1
Drug: Placebo — iv every 4 weeks for 24 weeks
  Arms: 2

SUMMARY:
This 2 arm study will compare the safety and efficacy, with regard to reduction of signs and symptoms, of tocilizumab versus placebo, both in combination with DMARDs, in patients with active rheumatoid arthritis who currently have an inadequate response to DMARD therapy. Patients will be randomized 2:1 to receive tocilizumab 8mg/kg iv or placebo iv every 4 weeks, in conjunction with stable DMARD therapy. The anticipated time on study treatment is 3-12 months, and the target sample size is 100-500 individuals.

ELIGIBILITY:
Inclusion Criteria:

* adult patients, 18-70 years of age;
* rheumatoid arthritis for >= 6 months;
* receiving permitted DMARDs, at a stable dose, for >= 8 weeks prior to baseline;
* current inadequate clinical response to DMARDs.

Exclusion Criteria:

* major surgery, including joint surgery, within 8 weeks before entering study, or planned major surgery within 6 months following randomization;
* rheumatic autoimmune disease or inflammatory joint disease other than rheumatoid arthritis;
* unsuccessful treatment with an anti-TNF agent;
* previous treatment with tocilizumab.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 209 (Actual)
Dates: Start 2008-10-31 (Actual); Primary Completion 2010-07-22 (Actual); Study Completion 2010-07-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (9):
- China (9):
  - Peking University People's Hospital, Beijing
  - Beijing Union Hospital, Beijing
  - General Hospital of Chinese PLA; Department of Hematology, Beijing
  - The Third Affiliated Hospital of Sun Yat-Sen University, Guangzhou
  - The 1st Affiliated Hospital of Harbin Medical University, Harbin
  - Qilu Hospital of Shandong University, Jinan
  - Renji Hospital Affiliated to Shanghai Jiao Tong University School of Medicine, Shanghai
  - Changhai Hospital of Shanghai, Shanghai
  - The First Affiliated Hospital of The Fourth Military Medical University (Xijing Hospital), Xi'an

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo + DMARDs: Participants received placebo intravenously (iv) every 4 weeks up to 24 weeks in combination with stable DMARD (disease modifying antirheumatic drugs) therapy
- Tocilizumab + DMARDs: Participants received tocilizumab 8 milligrams/kilogram (mg/kg) intravenously (iv) every 4 weeks up to 24 weeks in combination with stable DMARD (disease modifying antirheumatic drugs) therapy
Period: Overall Study
Arm/Group | Placebo + DMARDs | Tocilizumab + DMARDs
Started | 70 | 139
Completed | 65 | 135
Not Completed | 5 | 4
Not completed — Adverse Event | 1 | 3
Not completed — Withdrawal by Subject | 4 | 1

BASELINE CHARACTERISTICS:
Population: Intent-to-Treat (ITT) Population: The ITT population included all randomized participants who received at least one infusion of study treatment; Per Protocol (PP) Population: The PP population included all participants in the ITT population who adhered to the protocol.
Groups:
- Placebo + DMARDs: Participants received placebo intravenously every 4 weeks up to 24 weeks in combination with stable DMARD therapy
- Tocilizumab + DMARDs: Participants received tocilizumab 8 mg/kg intravenously every 4 weeks up to 24 weeks in combination with stable DMARD therapy
- Total: Total of all reporting groups
Arm/Group | Placebo + DMARDs | Tocilizumab + DMARDs | Total
Number analyzed (Participants) | 69 | 139 | 208
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.8 (11.68) | 46.8 (11.01) | 47.1 (11.22)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 55 | 120 | 175
  Male | 14 | 19 | 33

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With an American College of Rheumatology (ACR)20 Response at Week 24
Description: To achieve an ACR20 response required at least a 20% improvement, compared with baseline, in both (tender joints count)TJC and (swollen joints count) SJC, as well as in 3 out of 5 additional ACR core set variables: physician's global assessment of disease activity, participant's global assessment of disease activity, participant's assessment of pain, health assessment questionnaire disease index (HAQ-DI) and C-reactive protein (CRP). CRP was used primarily for the calculation of the ACR response; if missing, Erythrocyte Sedimentation Rate (ESR) was substituted. ITT sensitivity analysis was carried out using an alternative imputation method (last observation carried forward [LOCF]).
Time Frame: Week 24
Population: ITT Population
Measure: Number; unit: Percentage of Participants
Arm/Group | Placebo + DMARDs | Tocilizumab + DMARDs
Number analyzed (Participants) | 69 | 139
Percentage of Participants
  ITT Population | 24.6 | 69.8
  ITT Population (Sensitivity) | 24.6 | 73.4
Statistical Analysis 1: Comparison: Placebo + DMARDs vs Tocilizumab + DMARDs; Test type: Superiority or Other; p < 0.0001, Cochran-Mantel-Haenszel
Statistical Analysis 2: Comparison: Placebo + DMARDs vs Tocilizumab + DMARDs; Test type: Superiority or Other; p < 0.0001, Cochran-Mantel-Haenszel — ITT Population (Sensitivity)

2. Secondary Outcome: Percentage of Participants With ACR50 and ACR70 Responses at Week 24
Description: To achieve an ACR50 or ACR 70 response required at least a 50% or 70% improvement, compared with baseline in both TJC and SJC, as well as in 3 out of 5 additional ACR core set variables: physician's global assessment of disease activity, participant's global assessment of disease activity, participant's assessment of pain, HAQ-DI and CRP. CRP was used primarily for the calculation of the ACR response; if missing, ESR was substituted.
Time Frame: Week 24
Population: ITT Population
Measure: Number; unit: Percentage of Participants
Arm/Group | Placebo + DMARDs | Tocilizumab + DMARDs
Number analyzed (Participants) | 69 | 139
Percentage of Participants
  ACR 50 | 10.1 | 38.8
  ACR 70 | 2.9 | 12.9
Statistical Analysis 1: Comparison: Placebo + DMARDs vs Tocilizumab + DMARDs; Test type: Superiority or Other; p < 0.0001, Cochran-Mantel-Haenszel — Comparison of ACR 50 responders in placebo and Tocilizumab groups
Statistical Analysis 2: Comparison: Placebo + DMARDs vs Tocilizumab + DMARDs; Test type: Superiority or Other; p = 0.0345, Cochran-Mantel-Haenszel — Comparison of ACR 70 responders in placebo and Tocilizumab groups

3. Secondary Outcome: Number of Participants Who Received Escape Therapy
Description: Participants who did not achieve a 20% improvement from baseline in both SJC and TJC at week 16 could, if requested and deemed necessary by the investigator, receive escape therapy, comprising adjustment of the background DMARD dose and/or treatment with a different traditional DMARD.
Time Frame: 24 Weeks
Population: ITT Population
Measure: Number; unit: Number of participants
Arm/Group | Placebo + DMARDs | Tocilizumab + DMARDs
Number analyzed (Participants) | 69 | 139
Number of participants | 4 | 0

4. Secondary Outcome: Change in Tender and Swollen Joint Counts From Baseline to Week 24
Description: 68 joints were assessed for tenderness and joints were classified as tender/not tender giving a total possible tender joint count score of 0 to 68.
  66 joints were assessed for swelling and joints were classified as swollen/not swollen giving a total possible swollen joint count score of 0 to 66.
Time Frame: Baseline and Week 24
Population: ITT Population
Measure: Mean (Standard Deviation); unit: Joints
Arm/Group | Placebo + DMARDs | Tocilizumab + DMARDs
Number analyzed (Participants) | 69 | 139
Joints
  Swollen Joint Count | -4.5 (11.61) | -9.9 (9.26)
  Tender Joint Count | -6.2 (12.31) | -16.5 (12.06)
Statistical Analysis 1: Comparison: Placebo + DMARDs vs Tocilizumab + DMARDs; Placebo + DMARDs Vs Tocilizumab + DMARDs analysis for Swollen Joint Count; Test type: Superiority or Other; p < 0.0001, ANCOVA — p value was calculated using the difference between core set values of the two arms; Mean Difference (Final Values) = -4.7, 95% CI 2-sided [-6.6 to -2.8]
Statistical Analysis 2: Comparison: Placebo + DMARDs vs Tocilizumab + DMARDs; Placebo + DMARDs Vs Tocilizumab + DMARDs analysis for Tender Joint Count; Test type: Superiority or Other; p < 0.0001, ANCOVA — p value was calculated using the difference between core set values of the two arms; Mean Difference (Final Values) = -8.7, 95% CI 2-sided [-11.3 to -6.1]

5. Secondary Outcome: Change in Participant's Global Assessment of Disease Activity From Baseline to Week 24
Description: The participant's global assessment of disease activity is assessed on a 0 to 100 mm horizontal visual analogue scale (VAS) by the participant. The left-hand extreme of the line equals 0 mm, and is described as "no disease activity" (symptom-free and no arthritis symptoms) and the right-hand extreme equals 100 mm, as "maximum disease activity" (maximum arthritis disease activity). A negative change from Baseline indicated improvement.
Time Frame: Baseline and Week 24
Population: ITT Population
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Placebo + DMARDs | Tocilizumab + DMARDs
Number analyzed (Participants) | 65 | 132
mm | -8.7 (26.27) | -26.4 (24.69)
Statistical Analysis 1: Comparison: Placebo + DMARDs vs Tocilizumab + DMARDs; Test type: Superiority or Other; p < 0.0001, ANCOVA; Mean Difference (Final Values) = -19.1, 95% CI 2-sided [-25.3 to -12.9]

6. Secondary Outcome: Change in Physician's Global Assessment of Disease Activity From Baseline to Week 24
Description: The physician's global assessment of disease activity is assessed on a 0 to 100 mm horizontal VAS by the physician. The left-hand extreme of the line equals 0 mm, and is described as "no disease activity" (symptom-free and no arthritis symptoms) and the right-hand extreme equals 100 mm as "maximum disease activity" (maximum arthritis disease activity).
Time Frame: Baseline and Week 24
Population: ITT Population
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Placebo + DMARDs | Tocilizumab + DMARDs
Number analyzed (Participants) | 65 | 132
mm | -9.9 (22.61) | -29.1 (22.43)
Statistical Analysis 1: Comparison: Placebo + DMARDs vs Tocilizumab + DMARDs; Test type: Superiority or Other; p < 0.0001, ANCOVA; Mean Difference (Final Values) = -19.3, 95% CI 2-sided [-24.5 to -14.0]

7. Secondary Outcome: Change in Participant's Global Assessment of Pain From Baseline to Week 24
Description: The participants assessed their pain on a 0 to 100 mm VAS. The left-hand extreme of the line equals 0 mm, and is described as "no pain" and the right-hand extreme equals 100 mm as "unbearable pain". A negative change indicated improvement.
Time Frame: Baseline and Week 24
Population: ITT Population
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Placebo + DMARDs | Tocilizumab + DMARDs
Number analyzed (Participants) | 65 | 132
mm | -5.9 (23.97) | -23.5 (25.78)
Statistical Analysis 1: Comparison: Placebo + DMARDs vs Tocilizumab + DMARDs; Test type: Superiority or Other; p < 0.0001, ANCOVA; Mean Difference (Final Values) = -19.0, 95% CI 2-sided [-25.2 to -12.7]

8. Secondary Outcome: Change in C-Reactive Protein From Baseline to Week 24
Description: The serum concentration of CRP an acute phase inflammatory marker, is measured in milligrams/deciliter (mg/dL). A reduction in the level is considered an improvement.
Time Frame: Baseline and Week 24
Population: ITT Population
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Placebo + DMARDs | Tocilizumab + DMARDs
Number analyzed (Participants) | 65 | 132
mg/dL | -0.083 (2.310) | -1.865 (2.152)
Statistical Analysis 1: Comparison: Placebo + DMARDs vs Tocilizumab + DMARDs; Test type: Superiority or Other; p < 0.0001, ANCOVA; Mean Difference (Final Values) = -1.7384, 95% CI 2-sided [-2.1464 to -1.3303]

9. Secondary Outcome: Change in ESR From Baseline to Week 24
Description: The ESR was measured in mm/hour. A reduction in the level is considered an improvement.
Time Frame: Baseline and Week 24
Population: ITT Population
Measure: Mean (Standard Deviation); unit: mm/hour
Arm/Group | Placebo + DMARDs | Tocilizumab + DMARDs
Number analyzed (Participants) | 64 | 131
mm/hour | -4.4 (22.46) | -42.7 (26.23)
Statistical Analysis 1: Comparison: Placebo + DMARDs vs Tocilizumab + DMARDs; Test type: Superiority or Other; p < .0001, ANCOVA; Mean Difference (Final Values) = -39.2, 95% CI 2-sided [-44.7 to -33.7]

10. Secondary Outcome: Percentage of Participants With Low Disease Activity and in Clinical Remission
Description: DAS28 calculated from the number of swollen joints and tender joints using the 28-joint count, ESR and global health assessment (participant rated global assessment of disease activity using 10-mm VAS); DAS28 score ranged from 0 to 10, where higher scores correspond to greater disease activity. DAS28 less than or equal to (≤3.2) = low disease activity, DAS28 greater than (>)3.2 to 5.1 = moderate to high disease activity.
Time Frame: Baseline and Weeks 2, 4, 8, 12, 16, 20 and 24
Population: ITT Population; n=number of participants analyzed.
Measure: Number; unit: Percentage of Participants
Groups:
- Placebo+DMARD: Participants received placebo intravenously every 4 weeks up to 24 weeks in combination with stable DMARD therapy
Arm/Group | Placebo+DMARD | Tocilizumab + DMARDs
Number analyzed (Participants) | 69 | 139
Percentage of Participants
  Baseline Low Disease Activity (n= 69,139) | 0 | 0
  Baseline Remission (n=69, 139) | 0 | 0
  Baseline Remission first achieved (n=69, 139) | 0 | 0
  Week 2 Low Disease Activity (n= 67,138) | 0 | 2.2
  Week 2 Remission (n= 67,138) | 0 | 0.7
  Week 2 Remission first achieved (n= 67,138) | 0 | 0.7
  Week 4 Low Disease Activity (n= 67,139) | 0 | 12.9
  Week 4 Remission (n=67,139) | 0 | 5.0
  Week 4 Remission first achieved (n=67,139) | 0 | 5.0
  Week 8 Low Disease Activity (n= 67,139) | 1.5 | 24.5
  Week 8 Remission (n=67,139) | 0 | 12.9
  Week 8 Remission first achieved (n=67,139) | 0 | 8.6
  Week 12 Low Disease Activity (n=65,138) | 3.1 | 37.7
  Week 12 Remission (n=65,138) | 3.1 | 21.0
  Week 12 Remission first achieved (n=65,138) | 3.1 | 10.1
  Week 16 Low Disease Activity (n=65,136) | 6.2 | 39.0
  Week 16 Remission (n=65,136) | 1.5 | 24.3
  Week 16 Remission first achieved (n=65,136) | 1.5 | 7.4
  Week 20 Low Disease Activity (n=63,134) | 3.2 | 46.3
  Week 20 Remission (n=63,134) | 0 | 29.1
  Week 20 Remission first achieved (n=63,134) | 0 | 7.5
  Week 24 Low Disease Activity (n=64,131) | 4.7 | 46.6
  Week 24 Remission (n=64,131) | 3.1 | 30.5
  Week 24 Remission first achieved (n=64,131) | 1.6 | 4.6

11. Secondary Outcome: Change From Baseline to Week 24 in Functional Assessment of Chronic Illness Therapy (FACIT)-Fatigue Score
Description: FACIT-F is a 13-item questionnaire. Patients scored each item on a 5-point scale: 0 (Not at all) to 4 (Very much). The larger the participant's response to the questions (with the exception of 2 negatively stated), the greater the fatigue. For all questions, except for the 2 negatively stated ones, the code was reversed and a new score was calculated as (4 minus the participant's response). The sum of all responses resulted in the FACIT-Fatigue score for a total possible score of 0 (worse score) to 52 (better score). A higher score reflects an improvement in health status.
Time Frame: Baseline and Week 24
Population: ITT Population
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo + DMARDs | Tocilizumab + DMARDs
Number analyzed (Participants) | 61 | 132
units on a scale | 2.08 (7.684) | 6.51 (9.244)
Statistical Analysis 1: Comparison: Placebo + DMARDs vs Tocilizumab + DMARDs; Test type: Superiority or Other; p = 0.0003, ANCOVA; Mean Difference (Final Values) = 3.8, 95% CI 2-sided [1.8 to 5.9]

12. Secondary Outcome: Mean Rheumatoid Factor at Baseline and Week 24
Description: Rheumatoid factor (RF) is a disease characteristic and more than 85% of the participants studied were positive for the factor. These data are from patients who were RF positive. RF level was reported in international units/milliliter (IU/mL). A positive RF= >15 IU/mL.
Time Frame: Baseline and 24 Weeks
Population: ITT Population
Measure: Mean (Standard Deviation); unit: IU/mL
Arm/Group | Placebo + DMARDs | Tocilizumab + DMARDs
Number analyzed (Participants) | 61 | 125
IU/mL
  Baseline, n = 61, 125 | 179.5 (199.57) | 262.2 (360.39)
  Week 24, n = 57, 118 | 198.6 (277.06) | 204.6 (365.25)
Statistical Analysis 1: Comparison: Placebo + DMARDs vs Tocilizumab + DMARDs; Test type: Superiority or Other; p = 0.0599, ANCOVA; Mean Difference (Final Values) = -68.3, 95% CI 2-sided [-139.5 to 2.9]

13. Secondary Outcome: Change in Hemoglobin From Baseline to Week 24
Description: Levels of hemoglobin were determined in grams/liter (g/L)as a measure of anemia in participants
Time Frame: Baseline and 24 Weeks
Population: ITT Population
Measure: Mean (Standard Deviation); unit: g/L
Arm/Group | Placebo + DMARDs | Tocilizumab + DMARDs
Number analyzed (Participants) | 65 | 131
g/L | -1.0 (11.7) | 12.0 (14.1)
Statistical Analysis 1: Comparison: Placebo + DMARDs vs Tocilizumab + DMARDs; Test type: Superiority or Other; p < 0.0001, ANCOVA; Mean Difference (Final Values) = 12.956, 95% CI 2-sided [9.125 to 16.786]

14. Secondary Outcome: Change in Health Assessment Questionnaire - Disease Index (HAQ-DI) From Baseline to Week 24
Description: HAQ-DI is a self-completed participant questionnaire specific for RA. It consists of 20 questions referring to 8 domains: dressing/grooming, arising, eating, walking, hygiene, reach, grip; common daily activities. Each domain has at least 2 component questions. There are 4 possible responses for each component 0=without any difficulty 1=with some difficulty 2=with much difficulty 3=unable to do. The HAQ-DI is the sum of the scores, divided by the number of domains that have a score (in range 6-8) for a total possible score minimum/maximum 0 (best) to 3 (worst). A negative change from baseline indicated improvement.
Time Frame: Baseline and 24 Weeks
Population: ITT Population
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo + DMARDs | Tocilizumab + DMARDs
Number analyzed (Participants) | 65 | 132
units on a scale | -0.06 (0.522) | -0.52 (0.554)
Statistical Analysis 1: Comparison: Placebo + DMARDs vs Tocilizumab + DMARDs; Test type: Superiority or Other; p < 0.0001, ANCOVA; Mean Difference (Final Values) = -0.42, 95% CI 2-sided [-0.56 to -0.28]

15. Secondary Outcome: Percentage of Participants With ACR20 Response by First Week of Onset
Description: ACR 20 responses are summarized by first onset as a percentage of the total number of responders at week 24. The number of participants first achieving an ACR20 response at each time point is represented by treatment arm as a proportion of the total number of participants that had an ACR20 response at Week 24 using n as the denominator.
Time Frame: Weeks 2, 4, 8, 12, 16, 20, and 24
Population: ITT Population
Measure: Number; unit: Percentage of Participants
Arm/Group | Placebo + DMARDs | Tocilizumab + DMARDs
Number analyzed (Participants) | 17 | 97
Percentage of Participants
  First onset at Week 2 | 17.6 | 21.6
  First onset at Week 4 | 23.5 | 22.7
  First onset at Week 8 | 5.9 | 30.9
  First onset at Week 12 | 17.6 | 15.5
  First onset at Week 16 | 0 | 5.2
  First onset at Week 20 | 17.6 | 1.0
  First onset at Week 24 | 17.6 | 3.1

16. Secondary Outcome: Time to First Low Disease Activity
Description: Time to Low disease activity was calculated as the number of days from the first dose of drug administration to the date of first achievement of DAS28≤3.2.
Time Frame: Weeks 2, 4, 8, 12, 16, 20, and 24
Population: ITT Population
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Placebo + DMARDs | Tocilizumab + DMARDs
Number analyzed (Participants) | 69 | 139
Days | NA [172 to NA] — value not calculable due to insufficient events. | 139 [113 to 169]

17. Secondary Outcome: Time to First Remission
Description: Time to first Remission was calculated as the number of days from the date of first dose of study drug administration to the date of first achievement of DAS<2.6
Time Frame: Weeks 2, 4, 8, 12, 16, 20, and 24
Population: ITT Population
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Placebo + DMARDs | Tocilizumab + DMARDs
Number analyzed (Participants) | 69 | 139
Days | NA [NA to NA] — value not calculable due to insufficient events. | NA [169 to NA] — value not calculable due to insufficient events.

ADVERSE EVENTS:
Time Frame: Adverse events were monitored and recorded throughout the study.
Description: There are 70 participants randomized in Placebo+DMARDs group. Of these, 2 participants were excluded from safety population because one didn't receive any treatment while another received treatment but had no post-baseline safety assessment. Thus, a total of 68 participants were included in safety Population.
Arm/Group | Placebo + DMARDs | Tocilizumab + DMARDs
Serious Adverse Events (participants affected / at risk) | 4/68 | 1/139
Other Adverse Events (participants affected / at risk) | 19/68 | 59/139
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo + DMARDs (N=68) | Tocilizumab + DMARDs (N=139)
Abscess Limb (Infections and infestations) | 1 | 0
Herpes Zoster (Infections and infestations) | 1 | 0
Uterine Infection (Infections and infestations) | 1 | 0
Pyrexia (General disorders) | 1 | 0
Neutrophil Count Decreased (Investigations) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo + DMARDs (N=68) | Tocilizumab + DMARDs (N=139)
Upper respiratory tract infection (Infections and infestations) | 4 | 9
Nasopharyngitis (Infections and infestations) | 1 | 6
Influenza (Infections and infestations) | 3 | 1
Abscess limb (Infections and infestations) | 1 | 0
Cystitis (Infections and infestations) | 0 | 1
Helicobacter infection (Infections and infestations) | 1 | 0
Herpes zoster (Infections and infestations) | 1 | 0
Lung infection (Infections and infestations) | 0 | 1
Pharyngitis (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 0 | 1
Uterine infection (Infections and infestations) | 1 | 0
Alanine aminotransferase increased (Investigations) | 1 | 8
Neutrophil count decreased (Investigations) | 1 | 3
White blood cell count decreased (Investigations) | 0 | 4
Aspartate aminotransferase increased (Investigations) | 0 | 3
Transaminases increased (Investigations) | 1 | 1
Blood bilirubin unconjugated increased (Investigations) | 0 | 1
Blood creatinine increased (Investigations) | 1 | 0
Hepatic enzyme increased (Investigations) | 1 | 0
Aphthous stomatitis (Gastrointestinal disorders) | 0 | 3
Abdominal pain (Gastrointestinal disorders) | 1 | 1
Abdominal pain upper (Gastrointestinal disorders) | 1 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 2
Cheilitis (Gastrointestinal disorders) | 0 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 0
Gingival ulceration (Gastrointestinal disorders) | 0 | 1
Mouth ulceration (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 1 | 0
Stomatitis (Gastrointestinal disorders) | 0 | 1
Toothache (Gastrointestinal disorders) | 0 | 1
Leukopenia (Blood and lymphatic system disorders) | 0 | 9
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 2
Anaemia (Blood and lymphatic system disorders) | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 1 | 4
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 2
Skin disorder (Skin and subcutaneous tissue disorders) | 0 | 1
Pyrexia (General disorders) | 2 | 2
Fatigue (General disorders) | 1 | 0
Infusion related reaction (General disorders) | 0 | 1
Dizziness (Nervous system disorders) | 0 | 2
Neuropathy peripheral (Nervous system disorders) | 0 | 1
Tremor (Nervous system disorders) | 0 | 1
Dysfunctional uterine bleeding (Reproductive system and breast disorders) | 0 | 1
Dysmenorrhoea (Reproductive system and breast disorders) | 1 | 0
Menstruation irregular (Reproductive system and breast disorders) | 0 | 1
Uterine cervical erosion (Reproductive system and breast disorders) | 0 | 1
Hepatic function abnormal (Hepatobiliary disorders) | 0 | 3
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 1
Vision blurred (Eye disorders) | 0 | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Insomnia (Psychiatric disorders) | 2 | 0
Angina pectoris (Cardiac disorders) | 0 | 1
Hyperlipidaemia (Metabolism and nutrition disorders) | 0 | 1
Hypertension (Vascular disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The study being conducted under this agreement is part of the overall study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the study, but after the first publication or presentation that involves the overall study. Sponsor may request that confidential information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.